CLINICAL TRIAL: NCT04844593
Title: Use of Natural Language Processing (NLP) and Machine Learning (ML) for the Identification of Patients With Crohn's Disease (CD) and Complex Perianal Fistulas (CPF) and Their Characterization in Terms of Clinical and Demographic Characteristics. A Multicentre, Retrospective, NLP Based Study
Brief Title: A Study Using Artificial Intelligence to Identify Adults With Complex Perianal Fistulas Associated With Crohn's Disease
Acronym: INTUITION-CPF
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Darvadstrocel-5001
Record Dates: First submitted 2021-04-13; First posted 2021-04-14 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Crohn Disease; Rectal Fistula
Keywords: Drug Therapy
MeSH Terms: conditions — Crohn Disease; Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With CD: Participants with CD diagnosed with or without CPF will be identified from EMRs through medical language application program interface (API) software. The AI will apply NLP and machine learning to identify and analyse text information in EMRs and thereby, extract medical information. The data will be collected retrospectively from January 1st 2015 and December 31st 2021.

SUMMARY:
Natural Language Processing and machine learning are examples of artificial intelligence tools. This study will check if these tools correctly identify people with Crohn's disease with complex perianal fistulas from their medical records.

DETAILED DESCRIPTION:
This is a non-interventional, retrospective study of participants with CD and CPF in a clinical practice setting.

The study will enroll approximately 100 participants.

The study will have a retrospective data collection to select and analyze information from EMRs processed by an AI based analytics framework that uses machine learning and NLP methodologies.

All participants will be enrolled in one observational group.

• Participants with CD

This multi-center trial will be conducted in Spain. The overall duration of the study is approximately 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. CD participant diagnosed or not with CPF between January 1st 2015 and December 31st 2021.

Exclusion Criteria:

Not applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with CD diagnosed with or without CPF during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With CD and CPF Accurately Identified With the use of NLP and Medical Language (MEL) | Up to Month 36
  Percentage of participants will be measured in terms of accuracy and precision (sensitivity and specificity) of the "algorithm" used to identify participants with CPF associated with CD. Data obtained through the artificial intelligence (AI) technology will be compared with data obtained through traditional electronic data capture (EDC) and source data verification methods.

SECONDARY OUTCOMES:
Number of Participants With CD and CPF Characterized Using NLP and Machine Learning Techniques | Up to Month 36
  The following information at the moment of CPF diagnosis will be extracted from the electronical medical records (EMRs): age, gender, date of diagnosis of CPF, smoking status, date of diagnosis of CD, luminal disease characteristics (localization, behaviour and activity) at diagnosis, treatments (medical and surgical) established for luminal disease in the study period, treatments (medical and surgical) established for CPF since first occurrence, fistula characteristics at diagnosis: type of fistula (following American Gastroenterological Association [AGA] classification) number of fistula internal and external openings, fistula activity.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- Spain (3):
  - Hospital Universitario Son Espases, Palma, Balearic Islands
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Universitario Fundacion Alcorcon, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60774675688ad8001f42fba3